CLINICAL TRIAL: NCT07182266
Title: Perioperative Outcomes and Survival of Inflatable Video-Assisted Mediastinoscopic Transhiatal Esophagectomy for Selected Esophageal Cancer: A Comparative Study With Propensity-Score Matching Analysis
Brief Title: Perioperative Outcomes and Survival of Inflatable Video-Assisted Mediastinoscopic Transhiatal Esophagectomy for Selected Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2024-122R; 20ZR1411600 (Other Grant/Funding Number: Science and Technology Commission of Shanghai Municipality); SHDC2020CR4039 (Other Grant/Funding Number: Shanghai Hospital Development Center)
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Carcinoma
Keywords: esophageal carcinoma; mediastinoscopic; McKeown
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IVMTE: The patient was positioned supine. A 5-cm cervical incision was made along the anterior border of the left sternocleidomastoid muscle as the main surgical route. The skin and subcutaneous tissues were carefully incised in layers. The left recurrent laryngeal nerve (RLN) was identified and traced, followed by mobilization of the cervical esophagus. A lap protector was inserted into the left incision to create a closed cavity, and the mediastinum was insufflated with carbon dioxide at 8 mmHg. Three 5-mm trocars were used for the specialized retractor, LigaSure Maryland jaw sealer, and mediastinoscope. Then, the esophagus was dissected up to the level of the carina or the inferior pulmonary vein. During this process, mediastinal lymph nodes were also removed, including bilateral RLN, paraesophageal, tracheobronchial, and subcarinal nodes. If necessary, the incision was then extended to the right neck to facilitate the dissection of the right cervical lymph nodes.
- VME: traditional video-assisted McKeown esophagectomy

SUMMARY:
Perioperative and oncologic benefits of inflatable video-assisted mediastinoscopic transhiatal esophagectomy (IVMTE) are unclear. This retrospective study aimed to compare the differences in perioperative outcomes and survival between IVMTE and video-assisted McKeown esophagectomy (VME).

ELIGIBILITY:
Inclusion Criteria:

(I) primary esophageal cancer confirmed by endoscopic biopsy and (II) diagnosed resectable tumors based on positron emission tomography-computed tomography (PET-CT) according to the International Union Against Cancer Tumor, Node, Metastasis (TNM) Classification (8th edition)

Exclusion Criteria:

(I) presence of other advanced malignancies, (II) insufficient clinical data, or (III) postoperative follow-up of less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2021 to December 2023, patients with esophageal cancer who received IVMTE or VME were identified from the prospectively maintained esophageal cancer database at Zhongshan Hospital, Fudan University
Sampling Method: Non-Probability Sample
Enrollment: 1661 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Survival | within 2 years after surgery
  Disease-Free Survival, Overall Survival
Complication | perioperative
  follow the guidelines of the Esophageal Complications Consensus Group (ECCG) recommendations and Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
A data sharing plan is under consideration but must first be reviewed and approved by our ethics committee to ensure full compliance with participant confidentiality agreements.